CLINICAL TRIAL: NCT06862609
Title: Effect of the Quadro-Iliac Plane Block on Quality of Recovery Following Laparoscopic Inguinal Hernia Surgery: A Prospective, Randomized, Controlled, Double-Blind, Multicenter Study
Brief Title: QIPB in Inguinal Hernia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Muhammed Halit Satici, Specialist, M.D., Department of members Anesthesiology and Reanimation, Konya City Hospital, M.D, Konya City Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: QIPB İnguinal hernia
Record Dates: First submitted 2025-02-25; First posted 2025-03-06 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Other): All patients will receive IV paracetamol (1 g, 3×1) and IV tenoxicam (20 mg, 2×1). Rescue analgesia (IV tramadol 1 mg/kg) will be administered if Numerical rating scale scores are ≥3. IV ondansetron (4 mg) will be given for nausea and vomiting.
  Interventions: Other: Quadro iliac plane block
- Quadro iliac plane block (Active Comparator): All patients will receive IV paracetamol (1 g, 3×1) and IV tenoxicam (20 mg, 2×1). Rescue analgesia (IV tramadol 1 mg/kg) will be administered if Numerical rating scale scores are ≥3. IV ondansetron (4 mg) will be given for nausea and vomiting. Group Q patients will receive quadro iliac plane block in addition to standard analgesia.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Quadro iliac plane block — Patients in Group Q will be placed in the lateral position. A low-frequency convex transducer and a 100-mm block needle will be used. Following sterilization, the transducer will be placed parasagittally at the distal attachment of the quadratus lumborum muscle to the iliac crest. The iliac crest and quadratus lumborum muscle will be visualized, with the erector spinae muscle above and the psoas major muscle below. Using an in-plane technique, the needle will be directed toward the iliac crest. After confirmation with 5 mL of isotonic sodium chloride, 40 mL of 0.25% bupivacaine will be injected incrementally with intermittent aspiration.
  Arms: control group
Other: Control group — All patients will receive IV paracetamol (1 g, 3×1) and IV tenoxicam (20 mg, 2×1).
  Arms: Quadro iliac plane block

SUMMARY:
Inguinal hernia repair is one of the most commonly performed surgical procedures. It is generally performed under regional anesthesia techniques, such as local anesthesia, peripheral nerve blocks, or neuraxial anesthesia (spinal or epidural anesthesia), or under general anesthesia. Despite various available analgesic regimens, numerous studies have demonstrated that postoperative pain control remains inadequate. Opioids, nonsteroidal anti-inflammatory drugs, and analgesics are frequently used for postoperative pain management. However, these medications are associated with uncertain efficacy and undesirable side effects. Pain is a critical factor in the postoperative period, contributing to delayed ambulation and paralytic ileus, ultimately hindering early discharge.

DETAILED DESCRIPTION:
Inguinal hernia repair is one of the most commonly performed surgical procedures. It is generally performed under regional anesthesia techniques, such as local anesthesia, peripheral nerve blocks, or neuraxial anesthesia (spinal or epidural anesthesia), or under general anesthesia. Despite various available analgesic regimens, numerous studies have demonstrated that postoperative pain control remains inadequate. Opioids, nonsteroidal anti-inflammatory drugs, and analgesics are frequently used for postoperative pain management. However, these medications are associated with uncertain efficacy and undesirable side effects. Pain is a critical factor in the postoperative period, contributing to delayed ambulation and paralytic ileus, ultimately hindering early discharge. Recently, Tulgar and colleagues introduced a novel fascial plane block known as the "quadro-iliac plane block". Quadro-iliac plane block is performed within the quadro-iliac plane, located between the inner surface of the iliac crest and the posterior surface of the quadratus lumborum muscle. In their study, Tulgar et al. bilaterally injected 40 mL of methylene blue into the quadro-iliac plane. They observed widespread dye dispersion along the anterior and posterior surfaces of the quadratus lumborum muscle, transversalis fascia, ilioinguinal, iliohypogastric, subcostal, and genitofemoral nerves, as well as the lumbar plexus. Based on these findings, quadro-iliac plane block has been proposed as a potentially effective technique for managing acute or chronic pain in the lumbosacral, abdominal, and hip regions.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 years
* Undergoing elective,
* unilateral laparoscopic inguinal hernia repair
* Receiving general anesthesia

Exclusion Criteria:

* Patients who refuse to provide consent
* Patients with contraindications to regional anesthesia
* Patients with impaired consciousness
* Patients with coagulopathy
* Patients with infections at the block site
* Emergency cases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-03-23 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the QoR-15 score (0-150 point) at 24 hours postoperatively. | 24 hours
  The primary outcome is the QoR-15 score (0-150 point) at 24 hours postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Konya City Hospital, Konya, Turkey (Türkiye)